CLINICAL TRIAL: NCT02908815
Title: Investigating the Effect of Repetitive Transcranial Magnetic Stimulation (rTMS) as a Treatment for Alzheimer's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B2016:077
Record Dates: First submitted 2016-09-13; First posted 2016-09-21 (Estimated); Last update posted 2024-06-28 (Actual); Status verified 2021-02

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 4 weeks active treatment (Experimental): 4 weeks of rTMS active treatment applied using an active rTMS coil.
  Interventions: Device: rTMS active treatment
- 2 weeks active treatment (Experimental): 2 weeks of rTMS active treatment applied using an active rTMS coil.
  Interventions: Device: rTMS active treatment
- 4 weeks sham treatment (Sham Comparator): 4 weeks of rTMS sham treatment applied using a modified rTMS coil which does not stimulate the brain.
  Interventions: Device: rTMS sham treatment
- 2 weeks sham treatment (Sham Comparator): 2 weeks of rTMS sham treatment applied using a modified rTMS coil which does not stimulate the brain.
  Interventions: Device: rTMS sham treatment

INTERVENTIONS:
Device: rTMS active treatment — Repetitive Transcranial Magnetic Stimulation uses magnetic pulses to active neurons.
  Arms: 2 weeks active treatment; 4 weeks active treatment
Device: rTMS sham treatment — A fake treatment designed to mimic the sensations of rTMS
  Arms: 2 weeks sham treatment; 4 weeks sham treatment

SUMMARY:
The main objective of this study is to investigate the effects of repetitive Transcranial Magnetic Stimulation (rTMS) treatment on patients with probable early or moderate Alzheimer's disease.

DETAILED DESCRIPTION:
Upon meeting the inclusion criteria and providing informed consent, each participant will complete a series of cognitive assessments and rTMS treatments at the TMS Lab at Riverview Health Center (PE-450).

After enrollment, patients at each site will be assigned using stratified block randomization into either active or sham treatment arms with different duration of treatment (either 2 weeks or 4 weeks).

rTMS at frequency of 20 Hz will be used to stimulate the dorsolateral prefrontal cortex (DLPFC) of each patient in the real groups. Prior to the first treatment, and once per week during treatment, the patient's motor threshold will be measured using single pulses of TMS, noting the intensity necessary to cause a small twitch in the thumb finger. Then, the 70 mm cooled coil will be placed on the head at a location for optimal stimulation of the DLPFC at an intensity of 90-100% of the motor threshold. The 20 Hz rTMS treatment will incorporate 30 pulses per train, with 25 trains per side of the brain per session (total of 750 pulses per side per session). The trains will have a duration of 1.5 seconds, with an intertrain interval of 10 seconds. Each TMS treatment session will take approximately 10 to 25 minutes.

The DLPFC will be located on each patient using our Brainsight neuronavigation system from a reference MRI scan. If we cannot retrieve a valid previous clinical MRI scan or a valid ordered research MRI scan, a reference head model will approximate the patient's anatomy.

The treatments will be administered daily (5 days/week) either for 4 weeks or 2 weeks. The same protocol will also be used while doing sham stimulation.

To prevent un-blinding, the Magstim sham coil will be used; it provides the same sound and tactile sensory experience as those of the real coil, but it attenuates the strength of the induced electrical field in the brain well below the threshold required to stimulate neurons. In addition, during the treatment, only the designated research assistant and the patient will be present. It should also be noted that the only people who know the grouping are: the rTMS administrator (who also groups the patients) at each site and the sites' coordinator. The patients' grouping info will be in a secure folder in a locked cabinet to which only the rTMS administrator and the three sites coordinator will have the key.

Participants will be assessed six times during the study. This will occur at weeks 0, 3, 5, 13, 21, and 29 for the 4 week treatment groups, and weeks 0, 3, 5, 11, 19, and 27 for the 2 week treatment group. Each assessment will involve a set of nine assessment tools, including ADAS-Cog as the primary outcome measure and various other tasks and questionnaires to measure cognition, memory, caregiver burden, symptoms, and treatment tolerability.

For Winnipeg and Montreal sites only: The immediate effects (i.e. within 3 minutes) after participants receive the rTMS treatment will be assessed with a 1-minute semantic fluency test at four time points. This will occur at before and immediately after rTMS intervention in Week 1 and at weeks 5 and 13 for the 4 week treatment groups, and before and immediately after rTMS intervention in Week 1 and at weeks 5 and 11 for the 2 week treatment group.

Patients who are randomized to the sham treatment will be unblinded at the 6 month follow up and offered either 2-weeks or 4-weeks treatment; the patients and/or their family can choose the duration of treatment. As such, the 12 month assessment will be an unblinded follow up only of those initially randomised to one of the real groups (2-weeks or 4-weeks of treatment).

ELIGIBILITY:
Inclusion criteria:

* Individuals must have a MoCA score between 7 and 25, indicating mild cognitive impairment or dementia, a CDR score of 1-2, and a CSDD score of 18 or less.
* Participants must have probable early or moderate Alzheimer's disease as confirmed by their treating neurologist, geriatrician, or psychiatrist, and/or by the study doctors.
* Participants must be +55 years old.
* Participants must be taking a stable dose of an acetylcholinesterase inhibitor for at least 3 months prior to study entry with no plans to change medication for the duration of the study. Or if participants decide to stop taking their Alzheimer's disease related medication, they must wait a minimum of 6 weeks prior to the start of the intervention.

Exclusion criteria:

* Psychiatric conditions/disorders, or current neurological or medical disorders, other than AD, that could interfere with the subjects' cooperative participation (e.g. Severe agitation, prominent anxiety)
* Mental retardation
* Impaired visual and auditory acuity that confounds performance in cognitive tests
* Being diagnosed explicitly by other forms of dementia
* Confounding psychiatric disorders (e.g., schizophrenia, bipolar affective disorder) or current neurological, systemic, or medical disorders (e.g., liver disease, congestive heart failure, severe COPD) that may impair cognition and/or could affect attention span.
* Use of benzodiazepines or other hypnotics during the study and preceding two weeks
* Use of drugs with anticholinergic properties
* Pharmacological immunosuppression
* Participation in a clinical trial with any investigational agent within two weeks prior to study enrollment
* Current alcohol abuse
* History of epileptic seizures or epilepsy
* Contraindication for receiving TMS treatment according to a TMS questionnaire.
* Clinically significant abnormal laboratory findings which have not been approved by the Principal Investigator.
* Inability to adequately communicate in English in Manitoba and Australia sites and either English or French in Montreal site.
* Previous treatment with rTMS within the past 3 months
* A change in medication for AD, mood disorders, or pain during the study.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2022-08 (Actual); Study Completion 2022-08 (Actual)

PRIMARY OUTCOMES:
Alzheimer's Disease Assessment Scale-cognitive subscale (ADAS-Cog) change | Weeks 0 and 5
  Standard measure of cognitive symptoms, a popular tool that measures the severity of dementia symptoms. The primary outcome measure will be the change in the score from the baseline at 5 weeks.

SECONDARY OUTCOMES:
Stroop Test | Weeks 0, 3, 5, 11, 19, and 27 for the 2 week group and weeks 0, 3, 5, 13, 21, and 29 for the 4 week groups
  Measures a person's attention by having them read colour names when the colour of the text doesn't match.
Digit Span Test | Weeks 0, 3, 5, 11, 19, and 27 for the 2 week group and weeks 0, 3, 5, 13, 21, and 29 for the 4 week groups
  Memory test asking the participant to remember a sequence of numbers and repeat them back.
Verbal Fluency Test (VFT) | Weeks 0, 3, 5, 11, 19, and 27 for the 2 week group and weeks 0, 3, 5, 13, 21, and 29 for the 4 week groups
  Fluency test where the participant has to name as many words a possible that match a certain criteria.
Neuropsychiatric Inventory-Questionnaire (NPI-Q) | Weeks 0, 3, 5, 11, 19, and 27 for the 2 week group and weeks 0, 3, 5, 13, 21, and 29 for the 4 week groups
  Caregiver questionnaire that assesses severity of symptoms
Alzheimer's Disease Cooperative Study-Activities of Daily Living (ADCS-ADL) | Weeks 0, 3, 5, 11, 19, and 27 for the 2 week group and weeks 0, 3, 5, 13, 21, and 29 for the 4 week groups
  Caregiver questionnaire that assesses patient's ability to handle daily activities
Zarit Burden Interview (ZBI) | Weeks 0, 3, 5, 11, 19, and 27 for the 2 week group and weeks 0, 3, 5, 13, 21, and 29 for the 4 week groups
  Caregiver questionnaire that assesses the burden of the patient on the caregiver
Treatment Satisfaction Questionnaire for Medication (TSQM) | Weeks 3, 5, 11, 19, and 27 for the 2 week group and weeks 0, 3, 5, 13, 21, and 29 for the 4 week groups
  Assessment that asks directly if the participant is satisfied with the treatment
Alzheimer's Disease Assessment Scale-cognitive subscale (ADAS-Cog) effect over time | Weeks 0, 3, 11, 19, and 27 for the 2 week group and weeks 0, 3, 13, 21, and 29 for the 4 week groups
  Standard measure of cognitive symptoms, a popular tool that measures the severity of dementia symptoms.
Semantic Fluency Test (SFT) | Before and immediately after rTMS intervention in Week 1, at weeks 5 and 11 for the 2 week group and before and immediately after rTMS intervention in Week 1, at weeks 5, and 13 for the 4 week groups
  Fluency test where the participant has to name as many animals in 1 minute (Winnipeg and Montreal sites only)
Clinical Dementia Rating (CDR) sum of boxes | Week 27 for the 2 week group and week 29 for the 4 week group
  Assesses the severity of cognitive and functional decline related to Alzheimer's disease and other dementias

CONTACTS AND LOCATIONS:
Overall Officials: Zahra Moussavi, PhD, Principal Investigator — Department of Biomedical Engineering, University of Manitoba
Locations (3):
- Monash University, Melbourne, Victoria, Australia
- Canada (2):
  - Riverview Health Center, Winnipeg, Manitoba
  - McGill University, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
The data will be shared with two other institutes: McGill and Monash Universities, who are part of the same team.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 2016-12-01 till 2021-12-30
Access Criteria: Data are shared over a database that is only accessible by the sites of the study.

REFERENCES:
- [Derived] Moussavi Z, Uehara M, Rutherford G, Lithgow B, Millikin C, Wang X, Saha C, Mansouri B, Omelan C, Fellows L, Fitzgerald PB, Koski L. Repetitive transcranial magnetic stimulation as a treatment for Alzheimer's disease: A randomized placebo-controlled double-blind clinical trial. Neurotherapeutics. 2024 Apr;21(3):e00331. doi: 10.1016/j.neurot.2024.e00331. Epub 2024 Feb 14. PMID 38360452
- [Derived] Moussavi Z, Koski L, Fitzgerald PB, Millikin C, Lithgow B, Jafari-Jozani M, Wang X. Repeated Transcranial Magnetic Stimulation for Improving Cognition in Alzheimer Disease: Protocol for an Interim Analysis of a Randomized Controlled Trial. JMIR Res Protoc. 2021 Aug 9;10(8):e31183. doi: 10.2196/31183. PMID 34383681
- [Derived] Moussavi Z, Rutherford G, Lithgow B, Millikin C, Modirrousta M, Mansouri B, Wang X, Omelan C, Fellows L, Fitzgerald P, Koski L. Repeated Transcranial Magnetic Stimulation for Improving Cognition in Patients With Alzheimer Disease: Protocol for a Randomized, Double-Blind, Placebo-Controlled Trial. JMIR Res Protoc. 2021 Jan 8;10(1):e25144. doi: 10.2196/25144. PMID 33416500